CLINICAL TRIAL: NCT04517058
Title: The Influence of Comorbid Depression on the Prognosis of Patients With Newly-Diagnosed Epilepsy: A Prospective, Multi-center, Cohort Study
Brief Title: A Prospective Cohort Study on the Comorbid Depression in Patients With Newly-diagnosed Epilepsy
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Collaborators: Huashan Hospital (Other); Ruijin Hospital (Other); Shanghai 10th People's Hospital (Other); Shanghai 6th People's Hospital (Other); Shanghai East Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: NEWEpiDp
Record Dates: First submitted 2020-08-15; First posted 2020-08-18 (Actual); Last update posted 2021-12-28 (Actual); Status verified 2021-11

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- epilepsy patients with depression group: the score of HAMD-17>7
  Interventions: Other: psychology therapy
- epilepsy patients without depression group: the score of HAMD-17≤7

INTERVENTIONS:
Other: psychology therapy — If the symptoms are mild, patients will get the psychology therapy. If it's necessary according to patients' willings, patients will be given SSRIs antidepressant therapy.
  Other Names: SSRIs antidepressant drugs
  Groups: epilepsy patients with depression group

SUMMARY:
Epilepsy is a chronic brain disease with recurrent seizures and the comorbidity of psychiatric diseases are very common. The prevalence of depression in patients with refractory epilepsy is about 60%. However, the early diagnosis is usually difficult due to the unclear mechanism and untypical clinical symptoms, and there are no extremely effective treatments for depression in patients with epilepsy until now. In this prospective, multi-center, cohort study, we aim to investigate and screen two different types of depression ("cognitive" and "somatic") in patients with epilepsy by using the combination of regular moods evaluating scales and heart rate variability instrument. The intervening methods of combining transcranial direct current stimulation (tDCS) and serotonin re-uptake inhibitors (SSRIs) are used to treat the patients with comorbidity of epilepsy and depression.

DETAILED DESCRIPTION:
Epilepsy is a chronic brain disease with recurrent seizures and the comorbidity of psychiatric diseases are very common. The prevalence of depression in patients with refractory epilepsy is about 60%. However, the early diagnosis is usually difficult due to the unclear mechanism and untypical clinical symptoms, and there are no extremely effective treatments for depression in patients with epilepsy until now. In this prospective, multi-center, cohort study, we aim to investigate and screen two different types of depression ("cognitive" and "somatic") in patients with epilepsy by using the combination of regular moods evaluating scales and heart rate variability instrument. The intervening methods of combining transcranial direct current stimulation (tDCS) and serotonin re-uptake inhibitors (SSRIs) are used to treat the patients with comorbidity of epilepsy and depression. And resting-state functional MRI will be conducted in patients with the comorbidity of epilepsy and depression before and after the combing treatment of tDCS and SSRIs.

ELIGIBILITY:
Inclusion Criteria:

* meeting the definition of epilepsy according to the new definition issued by ILAE in 2014
* not using antidepressants
* acquiring informed consents

Exclusion Criteria:

* patients with severe psychiatric symptoms;
* progressive brain diseases
* malignant tumors
* severe cognitive declines

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: newly-diagnosed epilepsy
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2021-11-24 (Actual); Primary Completion 2023-09-30 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
the rate of seizure frequency | 12 months
  epilepsy diary

SECONDARY OUTCOMES:
the quality of life | 12 months
  scale

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Neurology, Zhongshan Hospital, Fudan University, Shanghai, China, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No